CLINICAL TRIAL: NCT07308145
Title: The Effect of Bruxism on Dynamic Balance in Desk Workers
Brief Title: The Effect of Bruxism on Balance
Status: Recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-250
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Orthopedic Physical Therapy; Bruxism
Keywords: Bruxism; Dynamic Balance; Desk Workers; Temporomandibular joint
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bruxism group: Bruxism group: Adults aged 18-50 years who have bruxism symptoms. Participants will undergo assessments of Masseter muscle stiffness, trigger points, quality of life, sleep quality, and dynamic balance.
  No experimental interventions are assigned.
- Non-bruxism group: Non-bruxism group: Adults aged 18-50 years those who do not have bruxism symptoms. Participants will undergo assessments of Masseter muscle stiffness, trigger points, quality of life, sleep quality, and dynamic balance.
  No experimental interventions are assigned.

SUMMARY:
This study will investigate the effect of bruxism on dynamic balance in desk-bound individuals. Participants will be divided into two groups based on whether they are diagnosed with bruxism or not. Dynamic balance and proprioception will be compared between individuals from each group.

DETAILED DESCRIPTION:
This observational study will include two groups: a bruxism group (n=27) and a Non-bruxism control group (n=27). At baseline, all participants will undergo the following assessments: Overall health-related quality of life 'Short Form 36 (SF-36)', Sleep quality (Pittsburgh Sleep Quality Index), Anxiety levels 'Beck Anxiety Inventory (BAI)', Head and jaw joint pain 'Fonseca Anamnestic Index (FAI)', Pain level 'Visual Analog Scale (VAS)', Perceived Stress Scale, Trigger Point Evaluation by a digital algometer, Assessment of dynamic balance by 'TecnoBody Prokin 252', Evaluation of the Masseter Muscle by 'Myoton PRO'. All procedures will be performed under standardized conditions with instructions and demonstrations provided to participants. Our study will evaluate the effect of bruxism on dynamic balance in desk-bound individuals and aims to compare the dynamic balance performance between individuals with and without bruxism.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years,
* Participants must be diagnosed with bruxism by a dentist,
* Voluntary participation and signing the informed consent form,
* The participant must have the cognitive capacity to communicate and understand instructions,
* Desk work hours must be at least 4 hours.

Exclusion Criteria:

* Unable to cooperate,
* Having active inflammatory arthritis,
* Having had hip or knee surgery within the last 3 months,
* Having a diagnosed psychiatric illness,
* Having dentofacial anomalies,
* Being pregnant,
* Having a physical or cognitive condition that would prevent completion of the given test protocols,
* Inability to comply with or cooperate with test procedures during the measurement period.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will include adults aged 18-50 years old, Participants will be divided into two groups based on whether they're diagnosed with bruxism or not. Each group will contain 27 individuals. All participants must be able to follow instructions clearly and complete the study assessments.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Short Form 36 (SF-36) | Single assessment during study visit (1 day)
  Quality of Life Scale/Short Form-36 (SF-36): SF-36 was developed by the Rand Corporation to obtain information about the health status of the individual. It was translated into Turkish by Koçyiğit and his colleagues, who conducted a validity and reliability study. It consists of eight sub-dimensions and 36 items. The sub-dimensions consist of physical function, social function, physical role difficulty, emotional state difficulty, mental health, energy/vitality, pain, and general perception of health. A score of "0" represents the worst health status, while "100" represents the best health status. Each sub-dimension is evaluated individually without calculating the total score.
Pittsburgh Sleep Quality Index | Single assessment during study visit (1 day)
  Pittsburgh Sleep Quality Index (PSQI): It is a 24-question scale developed by Buysse et al. in 1989 that evaluates sleep quality in the last month. A Turkish validity and reliability study was performed in 1996. The sum of the scores of seven components, subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, sleep medication use, and daytime dysfunction, gives the total score index. The total PSQI score ranges from 0 to 21; a score above 5 points indicates poor sleep quality; a score of 5 points or less indicates good sleep quality. The PSQI is one of the most commonly used scales for evaluating sleep quality. The validity of the use of this index in sleep disorders has been tested before, and it has been frequently used in studies on bruxism.
Beck Anxiety Inventory (BAI) | Single assessment during study visit (1 day)
  This scale's 21 items describe the most typical symptoms of anxiety disorders. It was developed to measure the intensity of anxiety symptoms in clinical populations. It asks respondents to indicate how much they have been affected by each symptom during the last week, on a scale from 0 (Not at all) to 3 (Severely - I could barely stand it). Total scores are the sum of all item scores, and range from 0 to 63; higher scores indicate higher anxiety. When this instrument was developed, the goal was to more easily discriminate between anxiety disorders and depressive disorders, whose symptoms frequently overlap on other assessment tools.
Fonseca Anamnestic Index | Single assessment during study visit (1 day)
  Fonseca Anamnestic Index (FAI): It was developed in 1994 by Fonseca et al. and consists of 10 questions investigating pain in the head and TMJ. Turkish validity and reliability of the test was performed by Kaynak et al. The questionnaire includes various questions about joint, head, and neck pain; joint movements; parafunctional habits; impaired occlusion; and emotional stress. Participants were asked to answer "Yes" , "Sometimes" , or "No" to each question, and TMD was classified as none, mild, moderate, or severe according to the total score.
Pain level-Visual Analog Scale (VAS) | Single assessment during study visit (1 day)
  Pain level-Visual Analog Scale: A visual analog scale (VAS) was used to assess the severity of pain related to bruxism. A VAS line was drawn on a 10 cm long horizontal line (0 = no pain and 10 = most intense pain), and the patient was asked to mark the pain intensity they perceived at rest, active use, and at night on this VAS line.
Trigger Point Evaluation | Single assessment during study visit (1 day)
  Trigger points in trapezius, masseter and temporalis muscles will be evaluated by algometre.
  Sudden reaction or vocal response of the patient with light pressure applied to this point and the presence of reflected pain in a region distant from this region indicated the presence of a trigger point (the minimum and maximum pressure sensitivity range varies from person to person, as it differs in sensitivity).
Perceived Stress Scale | Single assessment during study visit (1 day)
  Perceived Stress Scale: It was developed by Cohen, Kamarck, and Mermelstein in 1983 and consists of 14 items. Its Turkish validity and reliability was performed by Eskin et al., and this scale has been used in many studies on bruxism. The scale consists of two subdimensions: stress/discomfort perception and self-efficacy perception. Participants rate the stress they perceive on the scale as "0" never, "1" almost never, "2" sometimes, "3" often, and "4" very often. The stress level perceived by individuals is determined by summing the scores obtained from the items. A score between 0-56 points is obtained from the scale, and the higher the score, the higher the perceived stress level.
Measurement of dynamic balance | Single assessment during study visit (1 day)
  Balance assessments will be performed using Computerized Posturography (ProKin 252, Tecnobody, Dalmine, Italy), this device provides objectively measurable data for balance measurements.
  TecnoBody Prokin 252 will be used to measure and evaluate the patient's dinamik balance and proprioception levels in detail.
Evaluation of the Masseter's muscle stiffness | Single assessment during study visit (1 day)
  Masseter's muscle stiffness will be assessed with MyotonPRO. MyotonPRO (Muomeetria Ltd., Tallinn, Estonia) is a hand-held device used to quantify muscle stiffness. This device operates by generating a mechanical impulse on the skin overlying the muscle being assessed, followed by MyotonPRO measurements of the mechanical oscillations of muscles produced by the mechanical impulse. This method can determine the resistance of the muscle to deforming forces or muscle stiffness.

CONTACTS AND LOCATIONS:
Locations (1):
- İstinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
At this time, there is no finalized plan to share individual participant data (IPD). Data may contain sensitive personal information, and sharing will require additional ethical approvals and anonymization. Decisions regarding data sharing will be made after the study is completed.

REFERENCES:
- [Background] Chen Z, Shen Z, Ye X, Wu J, Wu H, Xu X. Association between Foot Posture Asymmetry and Static Stability in Patients with Knee Osteoarthritis: A Case-Control Study. Biomed Res Int. 2020 Jun 5;2020:1890917. doi: 10.1155/2020/1890917. eCollection 2020. PMID 32596282
- [Background] Silveira AM, Cericato GO, Meusel LDZV, Girotto LPDS, Bacchi A, Silva-Sousa YTC. Prevalence of temporomandibular disorders and associated factors: a population-based study in southern Brazil. Braz Oral Res. 2025 Sep 8;39:e092. doi: 10.1590/1807-3107bor-2025.vol39.092. eCollection 2025. PMID 40929410
- [Background] Divya M, Abinaya S, Alkousar Taz M, Manavalan N, Nivethitha L, Mooventhan A. Impact of yoga and naturopathy in a patient with unilateral Meniere's disease associated with pangastritis: A case report. J Bodyw Mov Ther. 2025 Dec;45:225-228. doi: 10.1016/j.jbmt.2025.08.032. Epub 2025 Aug 29. PMID 41316580
- [Background] Petzold Werle S, da Silveira J, de Azevedo Guimaraes AC. Effects of dance therapy on anxiety, stress, optimism and depressive symptoms in women undergoing breast cancer surgery: a randomized clinical trial. J Bodyw Mov Ther. 2025 Dec;45:516-523. doi: 10.1016/j.jbmt.2025.08.030. Epub 2025 Sep 4. PMID 41316614
- [Background] Huang D, Ke X, Jiang C, Song W, Feng J, Zhou H, Zhang R, Zhang A, Lan F. Effects of 12 weeks of Tai Chi on neuromuscular responses and postural control in elderly patients with sarcopenia: a randomized controlled trial. Front Neurol. 2023 Apr 28;14:1167957. doi: 10.3389/fneur.2023.1167957. eCollection 2023. PMID 37188307
- [Background] Luo W, Huang Z, Li H, Zhong T, Chen P, Min Y. Regulation of static and dynamic balance in healthy young adults: interactions between stance width and visual conditions. Front Bioeng Biotechnol. 2025 Jan 28;13:1538286. doi: 10.3389/fbioe.2025.1538286. eCollection 2025. PMID 39935603
- [Background] Luo W, Min Y, Chen P, Li H, Long Z, Sun J, Zhong T. Dual analysis of postural control in middle-aged and elderly patients with cervicogenic dizziness: Dynamic and static balance perspectives. Front Bioeng Biotechnol. 2025 Jul 22;13:1622648. doi: 10.3389/fbioe.2025.1622648. eCollection 2025. PMID 40766971
- [Background] Campos Lopez A, Estebanez-de-Miguel E, Camou Acedo T, Garcia-Pelagio KP, Albarova-Corral I, Malo Urries M, Villanueva-Melendez P. Reliability of myotonometry in the assessment of cervico-mandibular musculature: Inter/intra-examiner and inter/intra-session reliability study. Cranio. 2025 Jul 7:1-10. doi: 10.1080/08869634.2025.2528304. Online ahead of print. PMID 40620182
- [Background] Ucar I, Kararti C, Dadali Y, Ozudogru A, Okcu M. Masseter Muscle Thickness And Elasticity in Bruxism After Exercise Treatment: A Comparison Trial. J Manipulative Physiol Ther. 2022 May;45(4):282-289. doi: 10.1016/j.jmpt.2022.07.004. Epub 2022 Aug 31. PMID 36057478
- [Background] Galczynska-Rusin M, Pobudek-Radzikowska M, Gawriolek K, Czajka-Jakubowska A. Gender-Related Biomechanical Properties of Masseter Muscle among Patients with Self-Assessment of Bruxism: A Comparative Study. J Clin Med. 2022 Feb 5;11(3):845. doi: 10.3390/jcm11030845. PMID 35160297
- [Background] Yagci I, Tasdelen Y, Kivrak Y. Childhood Trauma, Quality of Life, Sleep Quality, Anxiety and Depression Levels in People with Bruxism. Noro Psikiyatr Ars. 2020 Mar 2;57(2):131-135. doi: 10.29399/npa.23617. eCollection 2020 Jun. PMID 32550779
- [Background] Machado NAG, Costa YM, Quevedo HM, Stuginski-Barbosa J, Valle CM, Bonjardim LR, Garib DG, Conti PCR. The association of self-reported awake bruxism with anxiety, depression, pain threshold at pressure, pain vigilance, and quality of life in patients undergoing orthodontic treatment. J Appl Oral Sci. 2020 Mar 27;28:e20190407. doi: 10.1590/1678-2019-0407. eCollection 2020. PMID 32236355
- [Background] Santos Miotto Amorim C, Firsoff EF, Vieira GF, Costa JR, Marques AP. Effectiveness of two physical therapy interventions, relative to dental treatment in individuals with bruxism: study protocol of a randomized clinical trial. Trials. 2014 Jan 7;15:8. doi: 10.1186/1745-6215-15-8. PMID 24398115
- [Background] Abasiyanik Z, Kopruluoglu M, Ucurum SG, Kahraman T, Kurt M, Keskin M, Kaya DO. Association Between Spinal Curvature and Mobility and Balance Abilities in Young Soccer Players. Percept Mot Skills. 2025 Oct;132(5):988-1004. doi: 10.1177/00315125251338539. Epub 2025 May 13. PMID 40364574
- [Background] Yu JF, Chang TT, Zhang ZJ. The Reliability of MyotonPRO in Assessing Masseter Muscle Stiffness and the Effect of Muscle Contraction. Med Sci Monit. 2020 Nov 2;26:e926578. doi: 10.12659/MSM.926578. PMID 33137025
- [Background] Kadioglu MB, Sezer M, Elbasan B. Effects of Manual Therapy and Home Exercise Treatment on Pain, Stress, Sleep, and Life Quality in Patients with Bruxism: A Randomized Clinical Trial. Medicina (Kaunas). 2024 Dec 4;60(12):2007. doi: 10.3390/medicina60122007. PMID 39768887
- [Background] Vazquez Morejon AJ, Vazquez-Morejon Jimenez R, Zanin GB. Beck Anxiety Inventory: psychometric characteristics in a sample from the clinical Spanish population. Span J Psychol. 2014 Oct 28;17:E76. doi: 10.1017/sjp.2014.76. PMID 26055653